CLINICAL TRIAL: NCT06838455
Title: Effectiveness of Therapeutic Exercises on Spinopelvic Mobility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Orthopedic Surgeon, Colorado Joint Replacement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2279537
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis (OA) of the Hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinopelvic Exercise (Experimental): Participants will complete a 15-20 min session of therapeutic exercises performed by patients with assistance of a pre-recorded video.
  Interventions: Other: Spinopelvic mobility exercise

INTERVENTIONS:
Other: Spinopelvic mobility exercise — Participants will complete a 15-20 min session of therapeutic exercises performed by patients with assistance of a pre-recorded video. The exercise regimen has been developed by the investigators of this study to incorporate exercises to increase a patient's spinopelvic mobility. Study staff that has been properly trained will be present to guide the patient through the exercise regimen and ensure the exercises are being performed accurately.

SUMMARY:
The purpose of this study is to examine the extent to which spinopelvic exercises may affect either sagittal spinal deformity or spinopelvic mobility and identifying patients at risk for hip instability following a total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-90 scheduled for total hip arthroplasty
2. Patients with primary hip osteoarthritis
3. Patients with or without history of prior spinal injections

Exclusion Criteria:

1. Patients undergoing revision total hip arthroplasty.
2. Patients with spinal fusion.
3. Patients who exercised prior to radiographic analysis.
4. Patients unable to complete imaging at the designated time of day.
5. Symptomatic contralateral hip osteoarthritis.
6. Patients unwilling or unable to perform therapeutic exercise program as instructed. This includes patients requiring use of assistive devices or who would be deemed unsafe to perform the exercises without a 1- or 2-person assist.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Spinopelvic radiographic measurements | Change from baseline to up to 1 hour after spinopelvic exercises same day.
  Spinopelvic parameter measurements on pre- and post-exercise radiographs including pelvic incidence, pelvic tilt, sacral slope and lumbar lordosis. All measurements are angles calculated in degrees.
Lumbar mobility | Change from baseline to up to 1 hour after spinopelvic exercises same day
  Calculated as the change in angle of lumbar lordosis between neutral standing and flexed-forward seated radiographs.
Spinopelvic mobility | Change from baseline to up to 1 hour after spinopelvic exercises same day
  Calculated as the change in angle of pelvic tilt between neutral standing and flexed-forward seated radiographs.
Patient risk classification for THA instability | Change from baseline to up to 1 hour after spinopelvic exercises same day
  Risk classification based on previously published risk factors for THA instability (lumbar stiffness, abnormal pelvic mobility, standing pelvic tilt greater than 13, sagittal spinal deformity)

SECONDARY OUTCOMES:
Oswestry Disability Index score | Baseline
  Patient reported outcome for pre-existing back pain and disability. The questionnaire is comprised of 10 sections, where each section is scored on a scale from 0 to 5 and summed. Higher score totals indicates worse disability.
Hip Society Score | Baseline
  Patient reported outcome, scored from 0 to 100. Higher scores indicate better outcomes.
Hip disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR) | Baseline
  Patient reported outcome, scored from 0 to 100. Higher scores indicate better outcomes.
The Veterans Rand 12-Item Health Survey scores (VR-12) | Baseline
  Patient reported outcome. Scores are reported as a Z-score that is based on the United States population average of 50. Higher scores indicate better outcomes.
Use of medication for hip/back pain | Baseline
  Assessed by standard of care questionnaire prior to the pre-operative visit with provider for a total hip replacement.
Severity of hip arthritis | Baseline
  Graded using Kellgren-Lawrence scale for osteoarthritis on AP radiographs. Grades are between 0-4, where 0 indicates an absence of osteoarthritis and a 4 indicates severe osteoarthritis.
Adverse events | Day 1
  Any adverse events sustained from therapeutic exercises

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Douglas, MD, Principal Investigator — Colorado Joint Replacement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dagneaux L, Marouby S, Maillot C, Canovas F, Riviere C. Dual mobility device reduces the risk of prosthetic hip instability for patients with degenerated spine: A case-control study. Orthop Traumatol Surg Res. 2019 May;105(3):461-466. doi: 10.1016/j.otsr.2018.12.003. Epub 2018 Dec 26. PMID 30594599
- [Background] Haws BE, Khechen B, Patel DV, Louie PK, Iyer S, Cardinal KL, Guntin JA, Singh K. Sagittal Imbalance Does Not Influence Cup Anteversion in Total Hip Arthroplasty Dislocations. Clin Spine Surg. 2019 Feb;32(1):E31-E36. doi: 10.1097/BSD.0000000000000712. PMID 30247184
- [Background] Buckland AJ, Abotsi EJ, Vasquez-Montes D, Ayres EW, Varlotta CG, Vigdorchik JM. Lumbar Spine Degeneration and Flatback Deformity Alter Sitting-Standing Spinopelvic Mechanics-Implications for Total Hip Arthroplasty. J Arthroplasty. 2020 Apr;35(4):1036-1041. doi: 10.1016/j.arth.2019.11.020. Epub 2019 Nov 22. PMID 31839349
- [Background] Buckland AJ, Fernandez L, Shimmin AJ, Bare JV, McMahon SJ, Vigdorchik JM. Effects of Sagittal Spinal Alignment on Postural Pelvic Mobility in Total Hip Arthroplasty Candidates. J Arthroplasty. 2019 Nov;34(11):2663-2668. doi: 10.1016/j.arth.2019.06.036. Epub 2019 Jun 22. PMID 31301908
- [Background] Lum ZC, Coury JG, Cohen JL, Dorr LD. The Current Knowledge on Spinopelvic Mobility. J Arthroplasty. 2018 Jan;33(1):291-296. doi: 10.1016/j.arth.2017.08.013. Epub 2017 Aug 24. PMID 28939031
- [Background] Murphy WS, Yun HH, Hayden B, Kowal JH, Murphy SB. The Safe Zone Range for Cup Anteversion Is Narrower Than for Inclination in THA. Clin Orthop Relat Res. 2018 Feb;476(2):325-335. doi: 10.1007/s11999.0000000000000051. PMID 29529664
- [Background] Abdel MP, von Roth P, Jennings MT, Hanssen AD, Pagnano MW. What Safe Zone? The Vast Majority of Dislocated THAs Are Within the Lewinnek Safe Zone for Acetabular Component Position. Clin Orthop Relat Res. 2016 Feb;474(2):386-91. doi: 10.1007/s11999-015-4432-5. PMID 26150264
- [Background] Esposito CI, Carroll KM, Sculco PK, Padgett DE, Jerabek SA, Mayman DJ. Total Hip Arthroplasty Patients With Fixed Spinopelvic Alignment Are at Higher Risk of Hip Dislocation. J Arthroplasty. 2018 May;33(5):1449-1454. doi: 10.1016/j.arth.2017.12.005. Epub 2017 Dec 13. PMID 29310920
- [Background] Tezuka T, Heckmann ND, Bodner RJ, Dorr LD. Functional Safe Zone Is Superior to the Lewinnek Safe Zone for Total Hip Arthroplasty: Why the Lewinnek Safe Zone Is Not Always Predictive of Stability. J Arthroplasty. 2019 Jan;34(1):3-8. doi: 10.1016/j.arth.2018.10.034. Epub 2018 Nov 2. PMID 30454867
- [Background] Ike H, Dorr LD, Trasolini N, Stefl M, McKnight B, Heckmann N. Spine-Pelvis-Hip Relationship in the Functioning of a Total Hip Replacement. J Bone Joint Surg Am. 2018 Sep 19;100(18):1606-1615. doi: 10.2106/JBJS.17.00403. No abstract available. PMID 30234627